CLINICAL TRIAL: NCT03785444
Title: Agreement in Relatives' Assessment in Standardized Questionnaires of Patients Who Have Been Admitted to Intensive Care Compared to Patients Who Have Not Been Admitted to Intensive Care (ASTON Study)
Brief Title: Comparison of Self-assessment vs. Assessment by Others of Critically Ill Patients
Acronym: ASTON
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other); Translationales intensivmedizinisches Forschungsnetzwerk Organdysfunktion (Unknown)
Responsible Party: Sponsor
Other Study IDs: ASTON
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Self-Assessment; Assessment, Self
Keywords: Assessment by others; Self-Assessment; Critically ill; Intensive care; standardized questionnaire; functional status; WHODAS; EQ5D; IADL; Barthel Score; SF-36; MoCA Blind
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Care Patients: Postoperative patients who have been admitted to intensive care
  Interventions: Other: WHODAS 2.0; Other: EQ5D; Other: IADL; Other: Barthel-Score; Other: SF-36; Other: MoCA Blind
- Non-Intensive Care Patients: Postoperative patients who have not been admitted to intensive care but to the normal ward
  Interventions: Other: WHODAS 2.0; Other: EQ5D; Other: IADL; Other: Barthel-Score; Other: SF-36; Other: MoCA Blind

INTERVENTIONS:
Other: WHODAS 2.0 — WHO Disability Score
Other: EQ5D — Health related quality of life measured with European Quality of Life 5 Dimensions 5 Level
Other: IADL — The Lawton Instrumental Activities of Daily Living
Other: Barthel-Score — Barthel Score of the patient
Other: SF-36 — Short Form Health 36
Other: MoCA Blind — Montreal Cognitive Assessment

SUMMARY:
We will test the results of standardized questionnaires for patients admitted to intensive care assessed by relatives/caregivers compared to the patient itself. Furthermore we will compare results with patients not admitted to intensive care.

ELIGIBILITY:
Inclusion Criteria:

* patient with a postoperative risk to be admitted to intensive care
* signed informed consent

Exclusion Criteria:

* patient who is not able to fill out the questionnaires alone and independent
* patient without relatives or a caregiver who could answer the assessment after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients with a high risk to be admitted to intensive care
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Agreement in assessment of ICU patients | 2 weeks before hospital admission
  Comparison of results of self-assessment versus assessment by others of standardized questionnaires of postoperative patients admitted to intensive care

SECONDARY OUTCOMES:
Agreement in assessment of ICU vs. non-ICU patients | 2 weeks before hospital admission
  Comparison of results of assessment of questionnaires of ICU patients vs. non-ICU patients
Agreement in assessment of non-ICU patients | 2 weeks before hospital admission
  Comparison of results of self-assessment versus assessment by others of standardized questionnaires of postoperative patients not admitted to intensive care but to the normal ward
Multivariate testing using the closeness of the relationship | 2 weeks before hospital admission
  It will be tested if the closeness of relationship patient - relative/caregiver changes the agreement, i.e. if the agreement is dependent or independent of the closeness of the relationship

OTHER OUTCOMES:
Definition of criteria which define an appropriate close relationship to receive a reliable test result | 2 weeks before hospital admission
  Test which closeness of relationship is sufficient to provide adequate test results compared with the patient's answers

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Technical University of Munich; Steffen Weber-Carstens, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar, School of Medicine, Technical University of Munich, Munich, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be made available to other researchers on reasonable request. A data share agreement will have to be signed by both parties.
  Examples of reasonable requests are:
  * a metaanalysis in the field
  * a research collaboration
  * rerun the analysis
  Data will only be provided for the purpose requested and may not be used otherwise without authorization/agreement.

REFERENCES:
- [Derived] Grunow JJ, Hartmann L, Ulm B, Maechler M, Blobner M, Seidenspinner K, Schoennagel L, Weber-Carstens S, Fuest K, Wollersheim T, Schaller SJ. Reliability of pre-admission patient-reported outcome measures postoperatively assessed via proxies: a prospective, multicenter observational study. Crit Care. 2025 May 19;29(1):200. doi: 10.1186/s13054-025-05431-6. PMID 40390142